CLINICAL TRIAL: NCT03738670
Title: Pain Evaluation After Treatment of Extra-spinal Bone Metastases With OsteoCOOL Radiofrequency (RF) Ablation System
Brief Title: Bipolar RFA of Painful Extra-spinal Bone Metastases
Acronym: PERFACOOL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 7010
Record Dates: First submitted 2018-11-05; First posted 2018-11-13 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Multi-metastatic Cancer
Keywords: Pain; Extra-spinal; RFA; Radiofrequency ablation; Bone metastases
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RFA (Experimental): Single-arm prospective observational study
  Interventions: Procedure: Percutaneous RFA

INTERVENTIONS:
Procedure: Percutaneous RFA — Single session percutaneous extra-spinal bone metastasis destruction to achieve pain relief

SUMMARY:
To evaluate the worst pain of cancer patients with painful extra-spinal bone metastases 1 month after bipolar radiofrequency ablation (RFA) performed with the Osteocool system.

ELIGIBILITY:
Inclusion Criteria:

* 1) Multi-metastatic cancer patients with at least one painful lytic bone metastasis
* 2) Target lesion should correspond to a specific radiologic finding
* 3) At least a moderate pain produce by target lesion (4 on a scale of 0 to 10 over the prior 24 hours with or without pain killers intake) assessed during selection evaluation
* 4) Patients 18 years old
* 5) Able to give written consent
* 6) Life expectancy 1 months
* 7) Patient affiliated to the National Health Insurance system

Exclusion Criteria:

1. Radiation therapy on the target tumor terminated < 3 weeks before treatment
2. Any contra-indication for the procedure as stated by the radiologist in terms of tumor size, proximity to neural/vascular structures making the procedure at unacceptable risk
3. Any contra-indication for the procedure as stated by the radiologist related to patient's condition (e.g. cardiac pacemakers) making the procedure at unacceptable risk
4. Impaired haemostasis
5. Concurrent participation in other experimental studies that could affect endpoints of this study
6. Contraindication to any form of sedation/anaesthesia
7. Signs of local/systemic infection identified before procedure, in accordance with standard care
8. Sclerotic metastases
9. Adults under guardianship
10. Patients under judicial protection
11. Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Percentage of responding patients reporting an improvement of at least 3 points on item 3 "the worst pain in the last 24 hours" of Brief Pain Inventory (BPI) questionnaire | 1 month

SECONDARY OUTCOMES:
Comparison of the mean scores of the items 3, 5, 9B and 8 of the BPI questionnaire between the baseline and 6-month follow-up | 6 months
Safety will be assessed according to SIR(11) / CTCAE classification | 6 months
Mean scores variation of the morphine milligram equivalents (MME) (based on patient consumption diary) between the baseline and 6-month follow-up. | 6 months
Percentage of responding patients defined by an improvement of at least 3 points on item 3 "the worst pain in the last 24 hours" of Brief Pain Inventory (BPI) questionnaire at 3 and 6 month follow-up. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Roberto CAZZATO, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- University Hospital, Strasbourg, france, Strasbourg, France